CLINICAL TRIAL: NCT00182065
Title: The Effect of Congestive Heart Failure on Functional and Cognitive Decline and Neuropsychiatric Symptoms in Residents of Long-term Care Facilities
Brief Title: Heart Failure, Functional and Cognitive Decline, and Psychiatric Symptoms in Nursing Home Patients
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 117947-BCA-CEBA-126289
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure, Congestive
Keywords: Heart failure; Functional decline; Cognitive impairment; Neuropsychiatric health; Longitudinal; Long-term care; Elderly
MeSH Terms: conditions — Heart Failure; Cognitive Dysfunction

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Heart failure is very common in the elderly, in whom it may lead to functional and intellectual problems. Functional problems include loss in the ability to perform basic tasks of daily living such as bathing or dressing. No studies have yet described the rate at which heart failure causes these problems to develop. This study aims to find out whether nursing home patients deteriorate more quickly with respect to function and intellect if they have heart failure. Participants will undergo a thorough health history and physical examination and will be followed every 3 months for up to a year. Over 30 nursing homes in Kitchener, Waterloo, Cambridge, and Hamilton, in South Central Ontario (Canada), are participating in this study. Every 3 months, participants will be reviewed with respect to function, intellect, mood and behaviours. Results between those with heart failure will be compared to those of people without heart failure. The results of this study will be used to plan further studies to see whether good treatment of heart failure can preserve function, intellect, and prevent depression and other mood problems.

DETAILED DESCRIPTION:
The prevalence of Heart Failure (HF) is rising, primarily among the elderly. HF has been diagnosed in 15 and 30% of elderly residents of long-term care facilities (LTCF). HF is associated with a high mortality rate and is the most common reason elderly persons are hospitalized. The economic impact of HF is substantial. Despite advances in the management of HF, the elderly are less likely to receive recommended therapies. This may reflect under-representation of the frail elderly in clinical trials of HF treatment. The elderly are more likely to experience adverse effects. In addition, HF trials have focused on mortality and hospitalization as outcome measures, which may be less relevant to the frail elderly who may be more concerned about preventing disability and preserving cognition.

Recent studies have demonstrated an association between functional decline, cognitive impairment and HF. Functional decline is defined as a loss in the ability to independently perform basic activities of self-care. In addition, patients with HF may be more likely to suffer from behavioural and psychological difficulties those without HF. The primary hypothesis of this study is that elderly residents of LTCF with a history of HF experience a more rapid rate of functional decline than residents without such a history. The secondary hypotheses are that elderly residents of LTCF with HF also experience a more rapid rate of cognitive decline and a greater burden of associated behavioural and psychological symptoms.

We propose to conduct a prospective cohort study in 25 LTCF in Hamilton, 9 LTCF in Kitchener-Waterloo, and 7 LTCF in Cambridge, all in Ontario. All newly admitted residents to these facilities will be considered for inclusion. Residents for whom consent cannot be obtained or who are not expected to survive more than eight weeks due to an underlying malignancy, end-stage neurological illness or other palliative diagnosis will be excluded. Approximately 600 patients will be recruited, 20% of which are expected to have a history of HF.

Residents for whom consent is obtained will be assessed by a research nurse. The assessment consists of a standardized history and physical examination, review of pertinent medical records, and an assessment of function (Barthel Index), cognition (MDS-COGS), and neuropsychiatric symptoms (Cohen-Mansfield Agitation Inventory and Neuropsychiatric Inventory). These measurements will be obtained at baseline and every three months thereafter for up to a year. The diagnosis of HF will be confirmed by two specialists using standard criteria. Residents with a history of HF will be compared to those without this history. Mortality, emergency room visits, acute hospitalizations, and falls will be measured.

Thus far, no studies have prospectively examined functional and cognitive decline in LTCF residents with HF. No studies have examined the relationship between HF and psychological and behavioural symptoms in these patients. As elderly residents of LTCF represent the frailest of the frail elderly, the results of this study are likely to be generalizable to the frail elderly in the community. We hope to apply the results of this study to future research aiming to determine whether treatment of HF can be optimized to reduce functional and cognitive decline in LTCF residents with HF, in order to preserve their independence and current level of disability as long as possible.

ELIGIBILITY:
Inclusion Criteria:

* All new residents to participating long-term care facilities
* Age 65 or over

Exclusion Criteria:

* Residing in any long-term care facility for more than 8 weeks
* Inability or refusal to obtain informed consent
* Palliative diagnosis and not expected to survive 6 weeks
* Residents admitted for respite care and expected to be returned to the community

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 586
Dates: Start 2004-03-01 (Actual); Primary Completion 2006-11-30 (Actual); Study Completion 2013-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George A Heckman, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Misiaszek B, Heckman GA, Merali F, Turpie ID, Patterson CJ, Flett N, McKelvie RS. Digoxin prescribing for heart failure in elderly residents of long-term care facilities. Can J Cardiol. 2005 Mar;21(3):281-6. PMID 15776118
- [Background] Heckman GA, Misiaszek B, Merali F, Turpie ID, Patterson CJ, Flett N, McKelvie RS. Management of heart failure in Canadian long-term care facilities. Can J Cardiol. 2004 Aug;20(10):963-9. PMID 15332144